CLINICAL TRIAL: NCT05946707
Title: Effects of Oxygen Supply on Hypoxic Pulmonary Vasoconstriction and Lung Collapse After Lung Isolation in Thoracic Surgery - a Prospective, Randomized Clinical Trial
Brief Title: Effects of Oxygen Supply After Lung Isolation in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1051/2023
Record Dates: First submitted 2023-05-25; First posted 2023-07-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation; Thoracic Surgery; One-Lung Ventilation
Keywords: Oxygen supply; Hypoxic pulmonary vasoconstriction; Lung collapse; Flow-controlled Ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: non-blinded, randomized, controlled trial
Who Masked: Participant
Masking Description: Study participants will be randomized after induction of general anesthesia and thus are not aware of the treatment arm, which solely differs at the time of lung isolation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high oxygen: decremental FiO2 titration (Active Comparator): Five minutes before lung isolation fraction of inspired oxygen will be increased to 1.0, representing the standard procedure for one-lung ventilation. 10, 20 and 30 minutes after OLV initiation paO2 obtained from arterial blood gas analysis will be measured and FiO2 titrated to achieve a paO2 of 75-120 mmHg.
  Interventions: Drug: liberal oxygen supply
- low oxygen: incremental FiO2 titration (Experimental): Before lung isolation fraction of inspired oxygen will be maintained as previously set to guarantee normoxia (SpO2 >92%). During OLV SpO2 will be continuously monitored and FiO2 adjusted to keep SpO2 >92%. Additionally after 10, 20 and 30 minutes after OLV initiation paO2 obtained from arterial blood gas analysis will be measured and FiO2 more precisely titrated to achieve a paO2 of 75-120 mmHg.
  Interventions: Drug: restrictive oxygen supply

INTERVENTIONS:
Drug: restrictive oxygen supply — Oxygen supply will be limited to guarantee normoxia at the beginning of OLV.
  Arms: low oxygen: incremental FiO2 titration
Drug: liberal oxygen supply — Oxygen supply will be maximized to 100% at the beginning of OLV
  Arms: high oxygen: decremental FiO2 titration

SUMMARY:
The goal of this randomized clinical trial is to compare a liberal versus restrictive oxygen supply (fraction of inspired oxygen, FiO2) strategy in patients scheduled for thoracic surgery requiring one-lung ventilation during lung isolation. The primary and secondary outcome parameters are:

* oxygenation of the blood after 30 minutes of one-lung ventilation, assessed by PaO2/FiO2 ratio
* time to lung collapse after start of one-lung ventilation

Participants in the control goup will receive an oxygen content of 100% before lung isolation, which will be subsequently decreased to achieve normoxia or mild hyperoxia (PaO2 of 75-120 mmHg).

The intervention group will receive the previous, during two-lung ventilation set, oxygen content and after lung isolation oxygen supply will be increased to secure adequate oxygenation of the blood (PaO2 75-120 mmHg) during one-lung ventilation.

The investigators hypothesize, that a higher fraction of inspired oxygen may impede hypoxic pulmonary vasoconstriction of the collapsed lung and thus decrease overall oxygenation performance during one-lung ventilation. Secondary endpoint will be the time to lung collapse, as a lower fraction of inspired oxygen and thus a higher nitrogen content may impede lung collapse.

DETAILED DESCRIPTION:
After anesthesia induction and securing the airway with a double lumen tracheal tube, the patient will be ventilated with pressure-controlled ventilation (PCV) and the following settings during two-lung ventilation (TLV): positive end-expiratory pressure of 5 cmH2O, peak pressure set to achieve a tidal volume of 6-8 ml/kg, respiratory rate set to achieve normocapnia, I:E ratio set to 1:1.5, FiO2 adjusted to achieve normoxia. After changing to lateral position, the patient will be randomized to one of the following group:

* Decremental FiO2 titration: FiO2 will be set to 1.0 five minutes before lung isolation and reduced consecutively during one-lung ventilation (OLV) according to paO2 measurement obtained from arterial blood gas samples to achieve normoxia (paO2 of 75-120 mmHg).
* Incremental FiO2 titration: FiO2 will be maintained to secure normoxia during the entire surgery. This means, that the previous FiO2 setting during two-lung ventilation will be continued and after OLV initiation the FiO2 has to be adjusted, to secure normoxia assessed by continuous SpO2 measurement (SpO2 of 92-96 %) and paO2 measurement obtained from arterial blood gas samples (paO2 of 75-120 mmHg).

During OLV the applied tidal volume will be reduced to 4-6 ml/kg by an appropriate adjustment of peak pressure, otherwise the ventilator settings will not be changed. After 30 minutes of OLV the intervention period ends and because in both groups oxygenation will be adjusted to achieve a PaO2 of 75-120 mmHg during OLV, the routine anesthetic regime of both groups will not differ in the further course of thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years
* Elective thoracic surgery requiring OLV
* American Society of Anesthesiologists physical status classification I-III
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Female subjects known to be pregnant
* Known participation in another interventional clinical trial
* Empyema evacuation or signs of pulmonary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
oxygenation of the blood | Primary outcome timepoint is defined at 30 minutes after start of OLV
  Oxygenation of the blood will be assessed by the paO2/FiO2 ratio and compared between groups.

SECONDARY OUTCOMES:
lung collapse | Lung collapse will be assessed and recorded as no collapse, partial collapse or complete collapse at 10, 20, 30 and 60 minutes after start of one-lung ventilation.
  Time to complete lung collapse will be recorded and compared between groups.
postoperative pulmonary complication | Follow-up will be completed after end of hospital stay or 30-days of hospital stay.
  Occurence of postoperative pulmonary complications will be assessed postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Spraider, MD, Principal Investigator — Medical University of Innsbruck, Department of Anesthesiology and Intensive Care Medicine
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No